CLINICAL TRIAL: NCT06138561
Title: Management of Cisplatin-Ineligible Patients With Metastatic Bladder Cancer and The Role of Geriatric Assessments
Status: Recruiting | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); EMD Serono (Industry)
Responsible Party: Principal Investigator, Joaquim Bellmunt, MD, Principal Investigator, Dana-Farber Cancer Institute
Other Study IDs: 23-478
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer; Metastatic Bladder Cancer; Unresectable Bladder Carcinoma; Urothelial Carcinoma
Keywords: Bladder Cancer; Metastatic Bladder Cancer; Unresectable Bladder Carcinoma; Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cisplatin-Ineligible Metastatic Bladder Cancer: Participants receiving standard of care non-cisplatin based therapy (carboplatin-based chemotherapy, enfortumab vedotin plus pembrolizumab or immunotherapy) and will complete study procedures as outlined below:
  * Baseline visit with questionnaires.
  * Complete surveys every 3 weeks by telephone or by in-office visit for 8 months.
  * Optional follow-up phone calls every 6 months for up to 3 years.
  Interventions: Behavioral: Geriatric-8 Survey; Behavioral: National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Bladder Symptom Index-18 (FBISI-18); Behavioral: Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®)

INTERVENTIONS:
Behavioral: Geriatric-8 Survey — A screening tool to evaluate frailty and at-risk participants by covering multiple domains that contribute to frailty, including mobility, functional status, pharmacologic burden, and underlying psychologic burden. A total score ranges from 0 to 17 with participants scoring > 14 points are more likely to be fit, or having a better health status, while those scoring 0 - 14 would benefit from further comprehensive geriatric assessment.
  Other Names: G8
Behavioral: National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Bladder Symptom Index-18 (FBISI-18) — Patient reported, sixteen question survey focused on evaluation of quality of life in patients with bladder cancer.
Behavioral: Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE®) — Patient-reported questionnaire that evaluates cancer-specific toxicity, developed based upon Common Terminology Criteria for Adverse Events.

SUMMARY:
The goal of this study is to better understand how to best treat participants with advanced bladder cancer who may not be able to tolerate all of the chemotherapy drugs that have been shown to be effective. In this study, investigators are assessing the role of the survey, the Geriatric-8, and its ability to predict outcomes in older participants undergoing cancer treatments. Additionally, investigators are evaluating the differential impact of treatments on quality of life in an older and at risk population.

DETAILED DESCRIPTION:
In this prospective, observational study, investigators are assessing the optimal approach to treating bladder cancer in older participants with other disease that might put the participants at additional risk from cancer-directed treatments. Investigators are specifically assessing the impact on adverse events, quality of life, and treatment outcomes. Additionally, investigators are assessing the role of the survey, the Geriatric-8, and its ability to predict outcomes in older participants.

The research study procedures include screening for eligibility and completing questionnaires.

Participation in this research study is expected to last for up to 8 months.

It is expected that about 180 people will take part in this research study.

The National Comprehensive Cancer Network and EMD Serono are supporting this research study by providing the necessary funds.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65-years-old (study will limit total enrollment of patients between ages 65-70 to 20% of the total study population)
* Unresectable or metastatic bladder cancer with histologically proven urothelial carcinoma. Any component of variant histology is allowed
* Cisplatin-ineligible as determined by the subject's primary oncologist
* Receiving treatment with chemotherapy (+/- immunotherapy maintenance), enfortumab vedotin-pembrolizumab combination therapy or immunotherapy alone
* Ability to understand and the willingness to sign a written informed consent document and to complete patient reported outcomes that will be in English or Spanish either alone or with assistance of study researcher or family

Exclusion Criteria:

* Subjects who elect to not undergo cancer-directed therapy
* Subjects obtaining their care outside of DFCI or DFCI affiliate sites
* Advanced cognitive impairment or inability to complete surveys
* Participants who are receiving any other investigational agents for this condition (if appropriate only).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Participants ≥65-years-old with metastatic or unresectable bladder cancer who are cisplatin-therapy ineligible.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life in frail and at-risk patients with advanced bladder cancer deemed cisplatin-ineligible | 8 months
  In frail and at-risk patients, as defined by geriatric-8 scores, will evaluate the difference in quality of life for participants receiving Carboplatin-based chemotherapy followed by immunotherapy maintenance versus Enfortumab Vedotin-Pembrolizumab. Quality of life will be measured by the National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Bladder Symptom Index-18 (NFBISI-18) version 2 questionnaire, a patient reported, eighteen question measure graded on a Likert scale.
Patient reported adverse events in frail and at-risk patients with advanced bladder cancer deemed cisplatin-ineligible | 8 months
  In frail and at-risk patients, as defined by geriatric-8 scores, will evaluate the difference in patient reported adverse events relevant to patients with bladder cancer between patients treated with Enfortumab Vedotin-Pembrolizumab vs. Carboplatin-based chemotherapy followed by immunotherapy maintenance. Patient reported adverse events will be assessed by the National Cancer Institute's Patient Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) questionnaire which will analyze 30 items, characterizing 16 symptomatic toxicities related treatment in terms of frequency, severity, interference (scoring from 0 to 4), and/or presence or absence (scoring 0 or 1).

SECONDARY OUTCOMES:
Frequency of acute care evaluations in patients with advanced bladder cancer deemed cisplatin-ineligible | 8 months
  In frail and at-risk patients as well as all study participants, will evaluate the difference in need for acute care evaluations in patients treated with Enfortumab Vedotin-Pembrolizumab versus Carboplatin-based chemotherapy followed by immunotherapy maintenance. Need for acute care evaluations will be are defined as the need for either hospitalizations or emergency department visits.
Frequency of treatment changes in patients with advanced bladder cancer deemed cisplatin ineligible | 8 months
  In frail and at-risk patients as well as all study participants, will evaluate the difference in need for treatment changes in patients treated with Enfortumab Vedotin-Pembrolizumab versus Carboplatin-based chemotherapy followed by immunotherapy maintenance. Treatment changes will be defined as dose adjustments, treatment disruption, or early treatment discontinuation.
Time to deterioration of quality of life in patients with advanced bladder cancer deemed cisplatin-ineligible | 8 months
  In frail and at-risk patients as well as all study participants, will evaluate the difference in time to deterioration of quality of life in patients treated with Enfortumab Vedotin-Pembrolizumab versus Carboplatin-based chemotherapy followed by immunotherapy maintenance. The time to deterioration of quality of life will be defined as a ≥ 3 point decrease from initial NFBISI-18 score on two consecutive evaluations (spaced 3 weeks apart) and will be analyzed using Kaplan-Meier estimates.
Overall survival in patients with advanced bladder cancer deemed cisplatin-ineligible | Up to 3 years
  In frail and at-risk patients as well as all study participants, will evaluate the difference in overall survival in patients treated with Enfortumab Vedotin-Pembrolizumab versus Carboplatin-based chemotherapy followed by immunotherapy maintenance. Overall survival will be defined as time from treatment initiation to death due to any cause or censored at date of last known alive. It will be analyzed using Kaplan-Meier estimates.
Geriatric-8 scores and acute care evaluations | 8 months
  In all study participants, will evaluate the association of geriatric-8 scores with need for acute care evaluations. Acute care evaluations are defined as the need for either hospitalizations or emergency department visits, which will be descriptively summarized.
Geriatric-8 scores and treatment changes | 8 months
  In all study participants, will evaluate the association of geriatric-8 scores with need for treatment changes.Treatment changes will be defined dose adjustments, treatment disruption, or early treatment discontinuation.
Geriatric-8 scores and time to deterioration of quality of life | 8 months
  In all study participants, will evaluate the association of geriatric-8 scores with time to deterioration of quality of life. Time to deterioration of quality of life will be defined as a ≥ 3 point decrease from initial NFBISI-18 score on two consecutive evaluations (spaced 3 weeks apart) and will be analyzed using Kaplan-Meier estimates according to G8 score.
Geriatric-8 scores and overall survival | Up to 3 years
  In all study participants, will evaluate the association of geriatric-8 scores with overall survival. Overall survival will be defined as time from treatment initiation to death due to any cause or censored at date of last known alive. It will be analyzed using Kaplan-Meier estimates according to G8 score

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Joaquim Bellmunt. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Background] Basch E, Reeve BB, Mitchell SA, Clauser SB, Minasian LM, Dueck AC, Mendoza TR, Hay J, Atkinson TM, Abernethy AP, Bruner DW, Cleeland CS, Sloan JA, Chilukuri R, Baumgartner P, Denicoff A, St Germain D, O'Mara AM, Chen A, Kelaghan J, Bennett AV, Sit L, Rogak L, Barz A, Paul DB, Schrag D. Development of the National Cancer Institute's patient-reported outcomes version of the common terminology criteria for adverse events (PRO-CTCAE). J Natl Cancer Inst. 2014 Sep 29;106(9):dju244. doi: 10.1093/jnci/dju244. Print 2014 Sep. PMID 25265940
- [Background] Taarnhoj GA, Lindberg H, Johansen C, Pappot H. Patient-reported outcomes item selection for bladder cancer patients in chemo- or immunotherapy. J Patient Rep Outcomes. 2019 Aug 22;3(1):56. doi: 10.1186/s41687-019-0141-2. PMID 31440865
- [Background] Peipert JD, Chang J, Li S, di Pietro A, Cislo P, Cappelleri JC, Cella D. Reliability, validity, and change thresholds of the NCCN/FACT Bladder Symptom Index (NFBlSI-18) in patients with advanced urothelial cancer. Cancer. 2024 Jan 1;130(1):31-40. doi: 10.1002/cncr.35025. Epub 2023 Oct 12. PMID 37823532
- [Background] Bellera CA, Rainfray M, Mathoulin-Pelissier S, Mertens C, Delva F, Fonck M, Soubeyran PL. Screening older cancer patients: first evaluation of the G-8 geriatric screening tool. Ann Oncol. 2012 Aug;23(8):2166-2172. doi: 10.1093/annonc/mdr587. Epub 2012 Jan 16. PMID 22250183